CLINICAL TRIAL: NCT00347451
Title: Optical Coherence Tomography Imaging of the Posterior Segment in High Myopia.
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Dr Laurence Lim, Singapore National Eye Centre
Other Study IDs: R415/10/2005
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Myopia; Maculopathy; Glaucoma
Keywords: myopia; optical coherence tomography
MeSH Terms: conditions — Myopia; Macular Degeneration; Glaucoma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The prevalence of myopia in East Asia and Singapore in particular is amongst the highest in the world, with estimates ranging from 30-70% of the general population. Up to 30% of these are high myopes. High myopia is associated with degenerative changes in the fundus. It may also be associated with vision-threatening complications such as macular holes. The pathogenesis of macular holes in high myopes is not completely understood but is postulated to include a combination of anterior vitreous traction and posterior staphyloma formation and axial elongation. These forces lead to degenerative changes at the macula, including foveal detachment and retinoschisis that precede the formation of lamellar or full thickness macular holes. These changes are difficult to detect either clinically or by conventional imaging such as ultrasound, making efforts to correct them in the early stages with surgery difficult. High myopia is also associated with a two- to threefold increase in risk of developing glaucoma. However, the diagnosis of glaucoma in high myopes is difficult as many of the pathological changes in the myopic eye mimic those seen in glaucoma. The myopic optic disc in particular is notoriously difficult to differentiate from the glaucomatous disc. Currently, the diagnosis is highly subjective, relying on observations of the clinical appearance of the disc or on disc photos.Optical coherence tomography (OCT) is an evolving technology that relies on time delays of reflected or backscattered light and interferometry to yield cross-sectional images of the retina and optic disc. The Stratus OCT is the latest model and has been demonstrated to be able to yield images with a resolution comparable to that of histology. It is thus potentially useful in assessing degenerative changes occurring in the myopic fundus, in evaluating the early changes preceding macular hole formation, and in providing objective measures of various disc parameters to aid in diagnosing glaucoma in high myopes. This study aims to recruit 150 healthy, young, ophthalmologically normal males from the SAF and to examine them with OCT. High myopes (≤-8D) will be selected and compared with a control group of low myopes. The performance of the OCT will be evaluated against current diagnostic methods.

DETAILED DESCRIPTION:
Primary AimThe aim of the study is to evaluate the retinal and macular topography, vitreomacular relationships and optic nerve head changes in highly myopic eyes of young adults. Specific aims include:1) To determine the prevalence of vitreo-macular traction and macular degenerations (macular thickening, detachments, schisis or lamellar holes) in asymptomatic, highly myopic young Asian males using OCT.2) To characterize and measure optic nerve head and peripapillary retinal nerve fibre layer changes in high myopia using OCT.3) To compare OCT findings with current methods of investigation and diagnosis

SubjectsSubjects will be drawn from in-service personnel as well as recruits awaiting enlistment. They will be identified based on their refraction through the SAF's computerized medical records system.Informed consent will be sought from the subjects before commencement. All subjects will be healthy young males and will be ophthalmologically normal apart from myopia. The main exclusion criteria are:1) Best corrected visual acuity <6/92) Previous intraocular surgery3) Intraocular pressure >21mmHg4) Gonioscopic findings of angle closure5) Clinical evidence of pseudo-exfoliation, uveitis or pigment dispersion syndrome, corneal or media opacities, retinal pathology or neurological diseases6) Family history in a first degree relative of glaucoma or other optic neuropathy.Excluded subjects will be replaced by the subject next-in-line in the cohort.ProcedureAll subjects identified will be examined at SNEC/SERI by one of the investigators. The assessment for each subject will include:1) Autorefraction performed with a non-accommodating target and recording of best corrected visual acuity. 2) Slit lamp examination, Goldmann applanation tonometry, gonioscopy, examination with a Goldmann three-mirror lens, and a dilated fundus examination with a 78 diopter fundus lens. Retinal findings are recorded in standard Amsler Dubois retinal diagrams. Grading of background myopic chorioretinal changes will be in accordance with the scheme proposed by Avila . 3) Axial length measurements. Ultrasound A scan is performed for each eye. Axial length is ascertained from the average of six consistent recordings. Care is taken to locate the fovea especially in cases with posterior staphyloma, by ensuring fixation of the A scan probe light. 4) Fundus photography with the Topcon camera. Stereoscopic disc photographs will also be taken for comparison with OCT scans of the optic nerve head.5) OCT using the Stratus OCTOCT measurements will be performed at one sitting by a trained technician. The commercially prescribed Optic Disc, RNFL and Macular Thickness scanning algorithms will be used. Each subject will fixate on an internal target presented by the computer where possible, or an external fixation target for cases unable to cooperate. Subjects will be encouraged to blink between the acquisition of each radial scan to minimize discomfort and minimize the effect of an irregular tear film or corneal desiccation on the tear film. Each scan will take approximately 2.5s, making for a total image acquisition time of less than a minute. The optic nerve head scan consists of six radial scans centered on the optic nerve head. The computer generated disc margin will be used as the reference for optic nerve head measurements. The macular thickness protocol uses six radial scans centered on the fovea. The retinal thickness is measured automatically as the distance between the vitreoretinal interface and the junction between the inner and outer segments of photoreceptors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adult males with myopia <-8D

Exclusion Criteria:

* Best corrected visual acuity <6/9
* Previous intraocular surgery
* Intraocular pressure >21mmHg
* Gonioscopic findings of angle closure
* Clinical evidence of pseudo-exfoliation, uveitis or pigment dispersion syndrome, corneal or media opacities, retinal pathology or neurological diseases
* Family history in a first degree relative of glaucoma or other optic neuropathy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Myopic subjects
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence S Lim, MBBS, Principal Investigator — Singapore National Eye Centre; Tin Aung, PhD, Study Director — Singapore National Eye Centre; Bobby C Cheng, FRCS, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

REFERENCES:
- [Background] Wong TY, Foster PJ, Hee J, Ng TP, Tielsch JM, Chew SJ, Johnson GJ, Seah SK. Prevalence and risk factors for refractive errors in adult Chinese in Singapore. Invest Ophthalmol Vis Sci. 2000 Aug;41(9):2486-94. PMID 10937558
- [Background] Tay MT, Au Eong KG, Ng CY, Lim MK. Myopia and educational attainment in 421,116 young Singaporean males. Ann Acad Med Singap. 1992 Nov;21(6):785-91. PMID 1295418
- [Background] Quek TP, Chua CG, Chong CS, Chong JH, Hey HW, Lee J, Lim YF, Saw SM. Prevalence of refractive errors in teenage high school students in Singapore. Ophthalmic Physiol Opt. 2004 Jan;24(1):47-55. doi: 10.1046/j.1475-1313.2003.00166.x. PMID 14687201
- [Background] Woo WW, Lim KA, Yang H, Lim XY, Liew F, Lee YS, Saw SM. Refractive errors in medical students in Singapore. Singapore Med J. 2004 Oct;45(10):470-4. PMID 15455167
- [Background] Phillips CI, Dobbie JG. Posterior Staphyloma and Retinal Detachment. Am J Ophthalmol. 1963 Feb;55:332-5. doi: 10.1016/0002-9394(63)92692-8. No abstract available. PMID 13943139
- [Background] Siam A. Macular hole with central retinal detachment in high myopia with posterior staphyloma. Br J Ophthalmol. 1969 Jan;53(1):62-3. doi: 10.1136/bjo.53.1.62. No abstract available. PMID 5775575
- [Background] Akiba J, Konno S, Yoshida A. Retinal detachment associated with a macular hole in severely myopic eyes. Am J Ophthalmol. 1999 Nov;128(5):654-5. doi: 10.1016/s0002-9394(99)00240-8. PMID 10577545
- [Background] Kishi S, Hagimura N, Shimizu K. The role of the premacular liquefied pocket and premacular vitreous cortex in idiopathic macular hole development. Am J Ophthalmol. 1996 Nov;122(5):622-8. doi: 10.1016/s0002-9394(14)70480-5. PMID 8909201
- [Background] Ripandelli G, Parisi V, Friberg TR, Coppe AM, Scassa C, Stirpe M. Retinal detachment associated with macular hole in high myopia: using the vitreous anatomy to optimize the surgical approach. Ophthalmology. 2004 Apr;111(4):726-31. doi: 10.1016/j.ophtha.2003.08.026. PMID 15051205
- [Background] Ishida S, Yamazaki K, Shinoda K, Kawashima S, Oguchi Y. Macular hole retinal detachment in highly myopic eyes: ultrastructure of surgically removed epiretinal membrane and clinicopathologic correlation. Retina. 2000;20(2):176-83. PMID 10783951
- [Background] Ichibe M, Yoshizawa T, Murakami K, Ohta M, Oya Y, Yamamoto S, Funaki S, Funaki H, Ozawa Y, Baba E, Abe H. Surgical management of retinal detachment associated with myopic macular hole: anatomic and functional status of the macula. Am J Ophthalmol. 2003 Aug;136(2):277-84. doi: 10.1016/s0002-9394(03)00186-7. PMID 12888050
- [Background] Hee MR, Puliafito CA, Duker JS, Reichel E, Coker JG, Wilkins JR, Schuman JS, Swanson EA, Fujimoto JG. Topography of diabetic macular edema with optical coherence tomography. Ophthalmology. 1998 Feb;105(2):360-70. doi: 10.1016/s0161-6420(98)93601-6. PMID 9479300
- [Background] Hee MR, Puliafito CA, Wong C, Duker JS, Reichel E, Schuman JS, Swanson EA, Fujimoto JG. Optical coherence tomography of macular holes. Ophthalmology. 1995 May;102(5):748-56. doi: 10.1016/s0161-6420(95)30959-1. PMID 7777274
- [Background] Azzolini C, Patelli F, Brancato R. Correlation between optical coherence tomography data and biomicroscopic interpretation of idiopathic macular hole. Am J Ophthalmol. 2001 Sep;132(3):348-55. doi: 10.1016/s0002-9394(01)01005-4. PMID 11530047
- [Background] Benhamou N, Massin P, Haouchine B, Erginay A, Gaudric A. Macular retinoschisis in highly myopic eyes. Am J Ophthalmol. 2002 Jun;133(6):794-800. doi: 10.1016/s0002-9394(02)01394-6. PMID 12036671
- [Background] Takano M, Kishi S. Foveal retinoschisis and retinal detachment in severely myopic eyes with posterior staphyloma. Am J Ophthalmol. 1999 Oct;128(4):472-6. doi: 10.1016/s0002-9394(99)00186-5. PMID 10577588
- [Background] Baba T, Ohno-Matsui K, Futagami S, Yoshida T, Yasuzumi K, Kojima A, Tokoro T, Mochizuki M. Prevalence and characteristics of foveal retinal detachment without macular hole in high myopia. Am J Ophthalmol. 2003 Mar;135(3):338-42. doi: 10.1016/s0002-9394(02)01937-2. PMID 12614751
- [Background] Panozzo G, Mercanti A. Optical coherence tomography findings in myopic traction maculopathy. Arch Ophthalmol. 2004 Oct;122(10):1455-60. doi: 10.1001/archopht.122.10.1455. PMID 15477456
- [Background] Rudnicka AR, Edgar DF. Automated static perimetry in myopes with peripapillary crescents--Part II. Ophthalmic Physiol Opt. 1996 Sep;16(5):416-29. PMID 8944186
- [Background] Aung T, Foster PJ, Seah SK, Chan SP, Lim WK, Wu HM, Lim AT, Lee LL, Chew SJ. Automated static perimetry: the influence of myopia and its method of correction. Ophthalmology. 2001 Feb;108(2):290-5. doi: 10.1016/s0161-6420(00)00497-8. PMID 11158801
- [Background] Jonas JB, Gusek GC, Naumann GO. Optic disk morphometry in high myopia. Graefes Arch Clin Exp Ophthalmol. 1988;226(6):587-90. doi: 10.1007/BF02169209. PMID 3209086
- [Background] Jonas JB, Dichtl A. Optic disc morphology in myopic primary open-angle glaucoma. Graefes Arch Clin Exp Ophthalmol. 1997 Oct;235(10):627-33. doi: 10.1007/BF00946938. PMID 9349946
- [Background] Dichtl A, Jonas JB, Naumann GO. Histomorphometry of the optic disc in highly myopic eyes with absolute secondary angle closure glaucoma. Br J Ophthalmol. 1998 Mar;82(3):286-9. doi: 10.1136/bjo.82.3.286. PMID 9602626
- [Background] Hyung SM, Kim DM, Hong C, Youn DH. Optic disc of the myopic eye: relationship between refractive errors and morphometric characteristics. Korean J Ophthalmol. 1992 Jun;6(1):32-5. doi: 10.3341/kjo.1992.6.1.32. PMID 1434043
- [Background] Schuman JS, Wollstein G, Farra T, Hertzmark E, Aydin A, Fujimoto JG, Paunescu LA. Comparison of optic nerve head measurements obtained by optical coherence tomography and confocal scanning laser ophthalmoscopy. Am J Ophthalmol. 2003 Apr;135(4):504-12. doi: 10.1016/s0002-9394(02)02093-7. PMID 12654368
- [Background] Mrugacz M, Bakunowicz-Lazarczyk A, Sredzinska-Kita D. Use of optical coherence tomography in myopia. J Pediatr Ophthalmol Strabismus. 2004 May-Jun;41(3):159-62. doi: 10.3928/0191-3913-20040501-08. PMID 15206601
- [Background] Avila MP, Weiter JJ, Jalkh AE, Trempe CL, Pruett RC, Schepens CL. Natural history of choroidal neovascularization in degenerative myopia. Ophthalmology. 1984 Dec;91(12):1573-81. doi: 10.1016/s0161-6420(84)34116-1. PMID 6084222
- [Background] Klein R, Klein BE, Wang Q, Moss SE. The epidemiology of epiretinal membranes. Trans Am Ophthalmol Soc. 1994;92:403-25; discussion 425-30. No abstract available. PMID 7886875
- [Background] Mitchell P, Smith W, Chey T, Wang JJ, Chang A. Prevalence and associations of epiretinal membranes. The Blue Mountains Eye Study, Australia. Ophthalmology. 1997 Jun;104(6):1033-40. doi: 10.1016/s0161-6420(97)30190-0. PMID 9186446
- [Background] Fraser-Bell S, Ying-Lai M, Klein R, Varma R; Los Angeles Latino Eye Study. Prevalence and associations of epiretinal membranes in latinos: the Los Angeles Latino Eye Study. Invest Ophthalmol Vis Sci. 2004 Jun;45(6):1732-6. doi: 10.1167/iovs.03-1295. PMID 15161833